CLINICAL TRIAL: NCT00299507
Title: Anecortave Acetate 15 mg Administered Every 3 Months Versus Anecortave Acetate 15 mg Administered Every 6 Months Versus Anecortave Acetate 30 mg Administered Every 6 Months in Patients With Exudative Age-Related Macular Degeneration (AMD)
Brief Title: Anecortave Acetate in Patients With Exudative Age-related Macular Degeneration (AMD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-04-59
Record Dates: First submitted 2006-03-03; First posted 2006-03-07 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2009-09

CONDITIONS: Macular Degeneration
Keywords: exudative AMD; age-related macular degeneration (AMD)
MeSH Terms: conditions — Macular Degeneration | interventions — anecortave acetate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 15 mg Anecortave Acetate, 3 month intervals (Experimental): Anecortave Acetate Sterile Suspension, 30 mg/mL, one 0.5 mL posterior juxtascleral depot injection at 3 month intervals (0, 3, 6, 9, 12, 15, 18 months).
  Interventions: Drug: Anecortave Acetate Sterile Suspension, 30 mg/mL
- 15 mg Anecortave Acetate, 6 month intervals (Experimental): Anecortave Acetate Sterile Suspension, 30 mg/mL, one 0.5 mL posterior juxtascleral depot injection at 6 month intervals (3, 9, 15, 21 months).
  Interventions: Drug: Anecortave Acetate Sterile Suspension, 30 mg/mL
- 30 mg Anecortave Acetate, 6 month intervals (Experimental): Anecortave Acetate Sterile Suspension, 60 mg/mL, one 0.5 mL posterior juxtascleral depot injection at 6 month intervals (3, 9, 15, 21 months).
  Interventions: Drug: Anecortave Acetate Sterile Suspension, 60 mg/mL
- Anecortave Acetate Vehicle (Sham Comparator): One 0.5 mL sham injection of Anecortave Acetate Vehicle at 6 month intervals (3, 9, 15, 21 months).
  Interventions: Other: Anecortave Acetate Vehicle

INTERVENTIONS:
Drug: Anecortave Acetate Sterile Suspension, 30 mg/mL — One 0.5 mL posterior juxtascleral depot injection at 3 or 6 month intervals
  Arms: 15 mg Anecortave Acetate, 3 month intervals; 15 mg Anecortave Acetate, 6 month intervals
Drug: Anecortave Acetate Sterile Suspension, 60 mg/mL — One 0.5 mL posterior juxtascleral depot injection at 6 month intervals
  Arms: 30 mg Anecortave Acetate, 6 month intervals
Other: Anecortave Acetate Vehicle — One 0.5 mL sham injection at 6 month intervals
  Arms: Anecortave Acetate Vehicle

SUMMARY:
The purpose of this study was to evaluate the effect of the dose concentration and administration frequency of Anecortave Acetate (AA) on visual acuity (VA) and lesion size when administered by posterior juxtascleral depot (PJD) every 3 months (AA 15 mg) or 6 months (AA 15 mg, AA 30 mg) in patients with exudative age-related macular degeneration (AMD).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of exudative AMD and a primary or recurrent (after laser photocoagulation) subfoveal choroidal neovascularization (CNV) lesion.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Less than 50 years of age.
* Other protocol-defined exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2005-03; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Mean change in best-corrected visual acuity (BCVA) at Month 12 from baseline | Month 12

SECONDARY OUTCOMES:
Mean change in lesion growth at Month 12 from baseline | Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Alcon Investigators, Principal Investigator — Alcon Research; Patricia Zilliox, Ph.D., Study Director — Alcon Research
Locations (1):
- Alcon Study Sites, Fort Worth, Texas, United States